CLINICAL TRIAL: NCT05240105
Title: Evaluation of the Suitability of the "Platform Model" as an Instrument for Staffing in Psychiatric and Psychosomatic Clinics (EPPIK) - Subproject Psychosomatics
Brief Title: Evaluation of the "Platform Model" for Staffing in Psychiatric and Psychosomatic Clinics
Acronym: EPPIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Deutsches Krankenhausinstitut (Unknown); DGPPN (Unknown); DGKJP (Unknown); DGPM (Unknown); Forum für Gesundheitswirtschaft gGmbH (Unknown)
Responsible Party: Principal Investigator, Simone Jennissen, Study coordinator, University Hospital Heidelberg
Other Study IDs: EPPIK
Record Dates: First submitted 2022-01-31; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Psychosomatic Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Departments for Psychosomatic Medicine at University Clinics: no study interventions, observational group
  Interventions: Other: no intervention, purely observational
- Clinics specialized in Psychosomatic Medicine: no study interventions, observational group
  Interventions: Other: no intervention, purely observational
- Departments for Psychosomatic Medicine at general hospitals: no study interventions, observational group
  Interventions: Other: no intervention, purely observational
- Departments for Psychosomatic Medicine at psychiatric hospitals: no study interventions, observational group
  Interventions: Other: no intervention, purely observational

INTERVENTIONS:
Other: no intervention, purely observational — There will be no interventions. The study is purely observational and investigates differences in naturally occuring treatments at these four types of departments for Psychosomatic Medicine.

SUMMARY:
This study aims to evaluate the so-called platform model and its suitability to determine staffing in hospitals for psychosomatic medicine and psychotherapy.

DETAILED DESCRIPTION:
The aim of the study is to test the suitability of a structural model (so-called platform model) developed by a working group of various scientific societies and professional associations for staffing in psychosomatic medicine and psychotherapy. For this purpose, in three steps (1.) the four treatment clusters developed in the platform model will be quantified and empirically validated on the basis of the therapeutic services provided in health care practice; (2.) the current staffing for the four treatment clusters will be described ("as-is analysis"); and (3.) prototypical therapy plans will be developed as a basis for estimating the target staffing requirements. On this basis, a target staffing estimate will be made for all professional groups.

For the study, a total of 80 psychosomatic clinics from Germany will be randomly selected, belonging in equal parts to the groups of psychosomatic university clinics, psychosomatic specialist hospitals, and psychosomatic departments in somatic or in psychiatric hospitals. In addition, 20 day clinics are included. In these clinics, the structural framework conditions including staffing will be surveyed and the routine documentation of therapy units will be evaluated by cluster analysis in order to empirically validate the presumed treatment clusters and to describe the necessary staffing requirements.

The empirical examination and validation of the platform model, including the four assumed treatment clusters, has the potential to positively influence care practice in the long term by adjusting staffing levels in psychosomatic clinics to actual care requirements.

ELIGIBILITY:
Inclusion Criteria for Clinics:

* belong to the predefined nationwide population of psychosomatic specialist clinics and departments
* randomly selected for inclusion in the study,
* the clinic management (head physician or comparable) agrees to participation in the study
* possibility of electronic recording of the qualified therapy units for all treating professional groups.

Inclusion Criteria for Patients:

* patient treated in one of the selected clinics on the corresponding ward or day clinic
* at least 18 years old

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nationwide German population of psychosomatic specialist clinics and departments at University hospitals, general hospitals, or psychiatric hospitals
Sampling Method: Probability Sample
Enrollment: 5961 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Administered Treatments | Week one of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week two of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week three of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week four of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week five of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week six of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week seven of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists
Administered Treatments | Week eight of treatment: assessment of administered treatment units
  units of psychotherapeutic treatment administered to each patient by physicians, psychologists, nurses, art therapists, social workers, and physiotherapists

SECONDARY OUTCOMES:
HONOS - Health of the Nation Outcome Scales | administered once per patient at week one of treatment
  measure of severity of mental illness

CONTACTS AND LOCATIONS:
Locations (1):
- Simone University Jennissen, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No